CLINICAL TRIAL: NCT01004549
Title: An Open-Label Evaluation of Degree of Accommodation in Pseudophakic Patients Bilaterally Implanted With Monofocal Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Innovative Medical (Industry)
Responsible Party: William Trattler MD, The Center for Excellence in Eye Care
Other Study IDs: Accomodation study
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Pseudophakia
Keywords: Patients who have previously undergone bilateral intraocular lens implantation
MeSH Terms: conditions — Pseudophakia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Bilateral intraocular lens implantation.

SUMMARY:
This study will determine the ability of three different intraocular lenses to accommodate in patients who have previously undergone bilateral intraocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 and older
* Patients must have undergone cataract surgery and have bilateral implants of the same model. The models eligible for inclusion include:

  * Crystalens
  * Crysalens HD
  * Tecnis One monofocal
* Patients must have a healthy cornea and macula
* Patients must have 20/25 or better best corrected vision
* Able to provide written informed consent

Exclusion Criteria:

* BCVA of less than 20/25
* On oral medications that could potentially block accommodation:

  * First generation antihistamines
  * Anticholinergic agents
  * Anti-psychotic medications
  * Antidepressant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Amplitude of accommodation on COAS and how it correlates with: spherical aberration on the COAS, pupil size at near as measured with COAS, spherical aberration on the topography, patient reported nead for spectacles for reading | one study visit

SECONDARY OUTCOMES:
Amplitude of accommodation on pushdown test - and how it compares to the COAS test results | one study visit

CONTACTS AND LOCATIONS:
Overall Officials: William Trattler, MD, Principal Investigator — The Center for Excellence in Eye Care
Locations (1):
- The Center for Excellence in Eye Care, Miami, Florida, United States